CLINICAL TRIAL: NCT00421278
Title: A Clinical Study to Evaluate the Efficacy and Safety of MK0633 in Patients With Atherosclerosis
Brief Title: The Effect of MK 0633 in Patients With Atherosclerosis (0633-008)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0633-008; MK0633-008; 2006_563
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — MK-0633 p-toluenesulfonate

ARMS (1):
- 1 (Experimental): Arm 1: Drug
  Interventions: Drug: MK0633

INTERVENTIONS:
Drug: MK0633 — Single dose MK0633 100mg po in the fed state administered during a 4-wk study.

SUMMARY:
A study to test the effects of study drug (MK 0633) on patients with Atherosclerotic disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with plaque in coronary or leg arteries, known as atherosclerosis or peripheral vascular disease
* Inflammatory marker found in your blood, known as hsCRP > 0.5 mg/L

Exclusion Criteria:

* Age < 40 or > 85
* Female
* Heart attack, coronary artery bypass, stroke or unstable angina in last 3 months
* Liver diseased or abnormalities
* HIV infection
* Lupus, rheumatoid arthritis, cancer <5 years

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-11; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of the drug, MK 0633, on an inflammatory marker in your blood that may affect the plaque in the arteries, know as atherosclerosis | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC